CLINICAL TRIAL: NCT02977364
Title: Phase I Trial to Investigate Safety and Tolerability Profile and Pharmacokinetics of C-met Kinase Inhibitor HS-10241 in Subjects With Advanced Solid Tumours
Brief Title: A Trial of C-met Kinase Inhibitor HS-10241 in Subjects With Advanced Solid Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10241-101
Record Dates: First submitted 2016-11-11; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma; Solid Tumor, Adult
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- HS-10241 100mg (Experimental): HS-10241 100mg daily
  Interventions: Drug: HS-10241
- HS-10241 200mg (Experimental): HS-10241 200mg daily
  Interventions: Drug: HS-10241
- HS-10241 400mg (Experimental): HS-10241 400mg daily
  Interventions: Drug: HS-10241
- HS-10241 600mg (Experimental): HS-10241 600mg daily
  Interventions: Drug: HS-10241
- HS-10241 800mg (Experimental): HS-10241 800mg daily
  Interventions: Drug: HS-10241
- HS-10241 1000mg (Experimental): HS-10241 1000mg daily
  Interventions: Drug: HS-10241

INTERVENTIONS:
Drug: HS-10241

SUMMARY:
To investigate safety, tolerability and pharmacokinetics of C-met Kinase Inhibitor HS-10241 in Subjects With Advanced Solid Tumours that are not eligible for conventional or intensive treatment. The dose of HS-10241 will be escalated to determine the dose limiting toxicity (DLT) and the maximum tolerated dose (MTD) of HS-10241 in advanced cancer patients. At the same time, pharmacokinetic characteristics and preliminary efficacy of HS-10241 will be observed in advanced cancer patients. To determine the recommended dosage regimen for phase II.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced or metastatic solid tumor for which standard therapy does not exist, has failed, or has been refused.
2. c-MET positive patients preferred in dose escalation phase; c-MET of patients must fulfill ICH++~+++ or FISH≥4 times in dose expansion phase.
3. Confirmed that there are at least 1 can be measured in accordance with the standard RECIST1.1 by CT or MRI.
4. 18 ~65 years of age.
5. ECOG performance status of 0~1.
6. Life expectancy of at least 3 months.
7. Recovered from toxicities of prior anti-cancer treatment to Grade 1 or less (except alopecia).
8. Acceptable hematologic status (without hematologic supports including hematopoietic factor, blood transfusion) defined below:

   * Absolute neutrophil count (ANC) ≥ 1500/μL
   * Platelet count ≥ 100000/μL
   * Hemoglobin ≥ 9.0 g/dL
9. Acceptable liver function defined below:

   * Total bilirubin ≤ 2 times upper limit of normal range (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times ULN; however, ≤ 5 times ULN in a subject who has liver metastases
10. Acceptable renal function defined below:

    * Serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance (by the Cockcroft-Gault formula) ≥ 60 mL/minutes
11. Acceptable coagulation status defined below:

    * Prothrombin time < 1.5 times ULN
    * Partial thrombin time < 1.5 times UL
12. HIV Ag/Ab(-).
13. HCV Ab(-);or HCV Ab(+) but HCV RNA(-).
14. HBsAg（-）and HBcAb（-）in dose escalation phase；HBV DNA<1×103copies/ml if HBsAg（+）or HBcAb（+）in dose expansion phase.
15. Ability to understand the purposes and risks of the trial and his/her informed consent using the human research ethics committee (HREC) approved informed consent form was obtained before the entering the trial.

Exclusion Criteria:

1. Treatment with other c-MET TKI( specific target or multi-target)；
2. Anti-cancer treatment with radiation therapy（not including non target lesions receiving palliative radiotherapy）, chemotherapy,hormonotherapy or surgery（small surgery, including the implantation of external equipment or fine needle aspiration, at least 7 days; diagnostic or palliative surgery, at least 14 days） within 4 weeks (6 weeks for nitrosoureas or Mitomycin C)prior to trial entry.
3. Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product
4. Cardiac disease with New York Heart Association (NYHA) Class III or IV, including congestive heart failure, myocardial infarction within 6 months prior to the trial entry, unstable arrhythmia, or symptomatic peripheral arterial vascular disease.
5. Symptomatic brain metastases or unstable brain metastases (notes: Patients with asymptomatic brain metastases previously treated for the study, but must be kept stable for at least 4 weeks and receive a stable dose of the drug)
6. Obvious neurological and mental disorder.
7. Other previous or concomitant tumors (except for the effective treatment of melanoma, cervical carcinoma in situ, ductal carcinoma in situ or malignant tumor after effective treatment, remission 3 years and considered to have been cured).
8. Active, uncontrolled bacterial, fungal infections, requiring systemic therapy.
9. Recent venous thrombosis (including deep vein thrombosis or pulmonary embolism within 0.5 year of trial entry)
10. History of organ allograft, autologous stem cell transplantation, or allogeneic stem cell transplantation.
11. Participation in an investigational drug or device trial within 4 weeks prior to the trial entry.
12. Anti-cancer treatment with radiation therapy, chemotherapy or immunotherapy within 4 weeks (6 weeks for nitrosoureas or Mitomycin C) prior to trial entry.
13. Major surgery, other than diagnostic surgery, within 4 weeks prior to the trial entry, without complete recovery
14. Taking a medication that is a moderate or strong inhibitor or inducer of CYP2C9; taking a medication that prolongs QT interval and has a risk of Torsades de Pointes .
15. Pregnant (positive serum beta human chorionic gonadotropin [β-HCG] test at Screening) or is currently breast-feeding, their partner anticipates becoming pregnant/impregnating during the trial or within 6 months after receiving the last dose of trial treatment.
16. Known drug abuse or alcohol abuse.
17. Concomitant disease or condition that could interfere with the conduct of the trial, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
MTD of HS-10241 based on the incidence of dose limiting toxicities | 4 weeks

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 12 months
Max concentration (Cmax) of HS-10241 | 4 weeks
Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 | 8 weeks
Incidence and intensity of Adverse Events according to Common Toxicity Criteria for AEs (CTCAE version 4.0) | 8 weeks
Area under the plasma concentration versus time curve (AUC) of HS-10241 | 4 weeks
Elimination half-life(T1/2) of HS-10241 | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No